CLINICAL TRIAL: NCT04643249
Title: A Phase I, Open-label, Fixed-sequence, Crossover, Drug-drug Interaction Study to Investigate the Inhibition Potential of KL1333 on CYP1A2, CYP2B6, CYP2C8, CYP2C9, CYP2C19, CYP2D6, and CYP3A4 in Healthy Subjects
Brief Title: Drug-drug Interaction Study of KL1333 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abliva AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KL1333 2020-103
Record Dates: First submitted 2020-11-13; First posted 2020-11-25 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Mitochondrial Disease
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Flurbiprofen; Dextromethorphan; Bupropion; Midazolam; Omeprazole; Caffeine; repaglinide

STUDY DESIGN:
Intervention Model Description: All subjects are treated in the same arm, but in a crossover manner.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): Daily treatment
  Interventions: Drug: KL1333; Drug: Flurbiprofen; Drug: Dextromethorphan; Drug: Bupropion; Drug: Midazolam injection; Drug: Omeprazole; Drug: Caffeine; Drug: Repaglinide

INTERVENTIONS:
Drug: KL1333 — Tablet
Drug: Flurbiprofen — Tablet
Drug: Dextromethorphan — Syrap
Drug: Bupropion — Tablet
Drug: Midazolam injection — solution for injection
  Other Names: Midazolam
Drug: Omeprazole — Capsule
Drug: Caffeine — Tablet or capsule
Drug: Repaglinide — Tablet

SUMMARY:
A Phase I, Open-label, Fixed-sequence, Crossover, Drug-drug Interaction Study to Investigate the Inhibition Potential of KL1333 on CYP1A2, CYP2B6, CYP2C8, CYP2C9, CYP2C19, CYP2D6, and CYP3A4 in Healthy Subjects

DETAILED DESCRIPTION:
This will be a Phase I, open-label, fixed-sequence, crossover study to investigate the effect of coadministration of KL1333 on the PK of repaglinide, caffeine, omeprazole, midazolam, bupropion, dextromethorphan, and flurbiprofen in healthy male and female subjects. Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the first dose administration. Subjects will be admitted into the clinical research unit (CRU) on Day -1 and be confined to the CRU until discharge on Day 19. Subjects will return to the CRU for a follow-up visit 5 to 7 days after the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 65 years of age, inclusive.
2. Weight ≥50 kg and body mass index between 18.0 and 32.0 kg/m2, inclusive.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhaemolytic hyperbilirubinaemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in as assessed by the investigator.
4. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception as detailed in Appendix 4.
5. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
6. Able to perform all protocol-specified assessments and comply with the study visit schedule.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator.
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, including KL1333 or its excipients, unless approved by the investigator.
3. History of gastroesophageal reflux disease, gastric erosions, peptic ulcer disease, or gastrointestinal bleeding episodes.
4. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs including cholecystectomy (uncomplicated appendectomy and hernia repair will be allowed).
5. History of malignancy of any organ system other than localised basal cell carcinoma of the skin, treated or untreated, within 5 years prior to screening, regardless of whether there is evidence of local recurrence or metastases.
6. History of clinically significant illness or surgery within 4 weeks prior to screening, as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Determination of the effect of KL1333 on the PK of repaglinide, caffeine, omeprazole, midazolam, bupropion, dextromethorphan, and flurbiprofen in healthy subjects. | day 14
  Area under the curve AUC

SECONDARY OUTCOMES:
evaluation of the single-dose PK of repaglinide, caffeine, omeprazole, midazolam, bupropion, dextromethorphan, and flurbiprofen administered alone and in the presence of KL1333 in healthy subjects | Day 14
  Area under the curve AUC
assessment of the safety and tolerability of KL1333 when coadministered with repaglinide, caffeine, omeprazole, midazolam, bupropion, dextromethorphan, and flurbiprofen in healthy subjects. | Day 14
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]).

CONTACTS AND LOCATIONS:
Locations (1):
- Volunteer recruitment center Covance Leeds Covance Leeds, Leeds, United Kingdom